CLINICAL TRIAL: NCT00499590
Title: A Phase 3, Randomized, Double-masked, Parallel-assignment Study of Intravitreal Bevasiranib Sodium, Administered Every 8 or 12 Weeks as Maintenance Therapy Following Three Injections of Lucentis® Compared With Lucentis® Monotherapy Every 4 Weeks in Patients With Exudative Age-Related Macular Degeneration (AMD).
Brief Title: Safety & Efficacy Study Evaluating the Combination of Bevasiranib & Lucentis Therapy in Wet AMD
Acronym: COBALT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACU301
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-09

CONDITIONS: Macular Degeneration
Keywords: AMD; Macular Degeneration; bevasiranib; COBALT study; age related macular degeneration; wet AMD; wet age related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — bevasiranib; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): Lucentis® (0.5mg) every 4 weeks.
  Interventions: Drug: ranibizumab
- B (Experimental): Bevasiranib (2.5mg) every 8 weeks beginning at week 12, after pre-treatment with 3 injections of Lucentis® and initial priming doses of bevasiranib at weeks 2 & 6.
  Interventions: Drug: bevasiranib
- C (Experimental): Bevasiranib (2.5mg) every 12 weeks beginning at week 12, after pre-treatment with 3 injections of Lucentis® and initial priming doses of bevasiranib at weeks 2 & 6.
  Interventions: Drug: bevasiranib

INTERVENTIONS:
Drug: bevasiranib — Bevasiranib (2.5mg) administered intravitreally every 8 or 12 weeks
  Arms: B; C
Drug: ranibizumab — Lucentis® (0.5 mg)administered intravitreally every 4 weeks.
  Other Names: Lucentis®
  Arms: A

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of bevasiranib given either every 8 weeks or every 12 weeks after an initial pre-treatment with 3 injections of Lucentis® (ranibizumab injection) compared to Lucentis® given every 4 weeks to people with wet AMD. Patients will be assigned at random (like tossing a coin) to receive one of three treatments options for 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be age 50 years or older
2. Patients must have predominantly classic, minimally classic or occult with no classic lesions secondary to Age Related Macular Degeneration.
3. The study eye must have ETDRS best corrected visual acuity of 69 to 24 letters (20/40 to 20/320 Snellen equivalent).
4. Patients must be willing and able to return for scheduled monthly follow-up visits for two-years.

Exclusion Criteria:

1. Prior pharmacologic treatment for AMD in the study (patients can not have previously received Avastin®/Lucentis®, Macugen®, or any other anti-VEGF agents, steroid treatments, PDT, radiation treatment, or any experimental therapies for AMD in the study eye)
2. Any intraocular surgery of the study eye within 12 weeks of screening
3. Previous posterior vitrectomy of the study eye
4. Advanced glaucoma or intraocular pressure above 22 mm Hg in the study eye despite treatment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2007-08; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis O'Shaughnessy, Ph.D., Study Director — Senior VP of Clincial Development
Locations (60):
- United States (55):
  - Retinal Consultants of Arizona (site 209), Phoenix, Arizona
  - Associated Retina Consultants (site 286), Phoenix, Arizona
  - Retina Centers PC (site 215), Tucson, Arizona
  - Eye Medical Center (site 287), Fresno, California
  - Northern California Retina Vitreous Associates (site 320), Mountain View, California
  - Retina Institute of California (site 207), Pasadena, California
  - Retina Consultants San Diego (site 232), Poway, California
  - Retinal Consultants Medical Group (site 289), Sacramento, California
  - Orange County Retina Medical Group (site 252), Santa Ana, California
  - Miramar Eye Specialists Medical Group (site 245), Ventura, California
  - The Eye Care Group, PC (site 315), Waterbury, Connecticut
  - Florida Eye Clinic (site 257), Altamonte Springs, Florida
  - Florida Eye Microsurgical Institute, Inc. (site 217), Boynton Beach, Florida
  - Retina Health Center (site 247), Fort Myers, Florida
  - National Ophthalmic Research Institute at Retina Consultants of SW Florida (site 270), Fort Myers, Florida
  - Magruder Eye Institute (site 264), Orlando, Florida
  - Southern Vitreoretinal Associates, PL (site 309), Tallahassee, Florida
  - University of South Florida Eye Institute (site 311), Tampa, Florida
  - Center for Retina and Macular Disease (site 293), Winter Haven, Florida
  - Southeast Retina Center (site 268), Augusta, Georgia
  - Midwest Eye Institute (site 253), Indianapolis, Indiana
  - Retina Associates, PA (site 295), Shawnee Mission, Kansas
  - Vitreo-Retinal Consultants & Surgeons, P.A. (site 274), Wichita, Kansas
  - Eye Centers of Louisville (site 251), Louisville, Kentucky
  - Retina Specialists (site 231), Towson, Maryland
  - Retina Associates St. Louis (site 300), Florissant, Missouri
  - Eye Foundation of Kansas City Truman Medical Center (site 272), Kansas City, Missouri
  - Retinal Consultants of Nevada (site 273), Las Vegas, Nevada
  - Eyesight Ophthalmic Services, PA (site 290), Portsmouth, New Hampshire
  - Delaware Valley Retina Associates (site 261), Lawrenceville, New Jersey
  - Retina-Vitreous Consultants (site 216), Livingston, New Jersey
  - Retina Associates of New Jersey (site 298), Teaneck, New Jersey
  - Capital Region Retina (site 316), Albany, New York
  - New York Eye & Ear Infirmary (site 272), New York, New York
  - Vitreous-Retina-Macula Consultants of New York (site 239), New York, New York
  - Carolina Eye Associates (site 308), Southern Pines, North Carolina
  - Retina Associates of Cleveland (site 228), Beachwood, Ohio
  - Cincinnati Eye Institute (site 285), Cincinnati, Ohio
  - Retina Associates of Cleveland, Inc. (site 219), Lakewood, Ohio
  - Retina-Vitreous Associates (site 266), Toledo, Ohio
  - Retina and Vitreous Center of Southern Oregon (site 271), Ashland, Oregon
  - Ophthalmology Associates of PA (site 297), Bala-Cynwyd, Pennsylvania
  - Palmetto Retina Center (site 275), West Columbia, South Carolina
  - Black Hills Regional Eye Institute (site 202), Rapid City, South Dakota
  - Southeastern Retina Associates, PC (Site 250), Knoxville, Tennessee
  - Retina Research Institute of Texas, L.L.C. (site 269), Abilene, Texas
  - Austin Retina Associates (site 304), Austin, Texas
  - Retina Research Center (site 204), Austin, Texas
  - University of Texas Medical Branch- Galveston (site 301, Galveston, Texas
  - Houston Eye Associates (site 321), Houston, Texas
  - Valley Retina Institue, PA (site 258), McAllen, Texas
  - Eye Care Associates of East Texas (site 282), Tyler, Texas
  - Rocky Mountain Retina Consultants (site 256), Salt Lake City, Utah
  - University of Utah, John A. Moran Eye Center (site 205), Salt Lake City, Utah
  - University of Virginia- Ophthalmology Dept. (site 254), Charlottesville, Virginia
- Canada (5):
  - Calgary Retina Consultants (site 318), Calgary, Alberta
  - Ivey Eye Institute (site 314), London, Ontario
  - Canadian Centre for Advanced Eye Therapeutics (site 291), Mississauga, Ontario
  - Sunnybrook Health Sciences Centre (site 305), Toronto, Ontario
  - Eye Centre Pasqua Hospital (site 299), Regina, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Groups:
- Lucentis®: Lucentis® (0.5mg) every 4 weeks.
  ranibizumab: Lucentis® (0.5 mg)administered intravitreally every 4 weeks.
- Bevasiranib 8 Weeks: Bevasiranib (2.5mg) every 8 weeks beginning at week 12, after pre-treatment with 3 injections of Lucentis® and initial priming doses of bevasiranib at weeks 2 & 6.
  bevasiranib: Bevasiranib (2.5mg) administered intravitreally every 8 or 12 weeks
- Bevasiranib 12 Weeks: Bevasiranib (2.5mg) every 12 weeks beginning at week 12, after pre-treatment with 3 injections of Lucentis® and initial priming doses of bevasiranib at weeks 2 & 6.
  bevasiranib: Bevasiranib (2.5mg) administered intravitreally every 8 or 12 weeks
Period: Overall Study
Arm/Group | Lucentis® | Bevasiranib 8 Weeks | Bevasiranib 12 Weeks
Started | 113 | 112 | 113
Completed | 0 | 0 | 0
Not Completed | 113 | 112 | 113
Not completed — Study Terminated | 112 | 112 | 112
Not completed — Not treated | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lucentis: Lucentis® (0.5mg) every 4 weeks.
  ranibizumab: Lucentis® (0.5 mg)administered intravitreally every 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Lucentis | Bevasiranib 8 Weeks | Bevasiranib 12 Weeks | Total
Number analyzed (Participants) | 113 | 112 | 113 | 338
Age, Continuous [Mean (Full Range); unit: years] | 77.6 [56 to 90] | 77.2 [52 to 95] | 78.3 [57 to 94] | 77.7 [52 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 72 | 59 | 211
  Male | 33 | 40 | 54 | 127
Region of Enrollment [Number; unit: participants]
  United States | 61 | 59 | 64 | 184
  Austria | 4 | 5 | 4 | 13
  Canada | 8 | 10 | 5 | 23
  France | 22 | 24 | 20 | 66
  Israel | 9 | 7 | 6 | 22
  Italy | 5 | 2 | 2 | 9
  Portugal | 3 | 3 | 5 | 11
  Spain | 1 | 2 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: avoidance of 3 or more lines of vision loss
Time Frame: week 60
Population: Zero participants analyzed due to early termination of the study.
Arm/Group | Lucentis® | Bevasiranib 8 Weeks | Bevasiranib 12 Weeks
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Need for Rescue Therapy, Time to Rescue Therapy, and Number of Patients With a 3 or More Line Gain in Vision
Time Frame: Week 60
Population: Zero participants analyzed due to early termination of the study.
Arm/Group | Lucentis | Bevasiranib 8 Weeks | Bevasiranib 12 Weeks
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Study was terminated early. Adverse events collected from first enrolled until study terminated, approximately 20 months.
Description: Safety population included randomized participants who received at least one treatment. Therefore the number of participants analyzed in the Lucentis and Bevasiranib 12 Weeks is one participant fewer than the number of participants randomized.
Arm/Group | Lucentis | Bevasiranib 8 Weeks | Bevasiranib 12 Weeks
Serious Adverse Events (participants affected / at risk) | 26/112 | 28/112 | 33/112
Other Adverse Events (participants affected / at risk) | 71/112 | 85/112 | 96/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lucentis (N=112) | Bevasiranib 8 Weeks (N=112) | Bevasiranib 12 Weeks (N=112)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Visual acuity decreased (Eye disorders) | 5 | 7 | 10
Endophthalmitis (Eye disorders) | 0 | 4 | 1
Uveitis (Eye disorders) | 0 | 1 | 2
Vitritis (Eye disorders) | 0 | 3 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 2
Cataract (Eye disorders) | 0 | 1 | 0
Corneal oedema (Eye disorders) | 1 | 0 | 0
Hyphaema (Eye disorders) | 0 | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 0 | 1
Macular degeneration (Eye disorders) | 0 | 0 | 1
Punctate keratitis (Eye disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Keratitis herpetic (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Heart rate irregular (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 2
Transient ischemia attack (Nervous system disorders) | 0 | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Dementia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lucentis (N=112) | Bevasiranib 8 Weeks (N=112) | Bevasiranib 12 Weeks (N=112)
Retinal haemorrhage (Eye disorders) | 11 | 16 | 22
Visual acuity reduced (Eye disorders) | 4 | 8 | 12
Conjunctival haemorrhage (Eye disorders) | 10 | 9 | 13
Vitreous detachment (Eye disorders) | 8 | 11 | 10
Vitreous floaters (Eye disorders) | 9 | 10 | 8
Eye pain (Eye disorders) | 6 | 7 | 12
Macular degeneration (Eye disorders) | 5 | 7 | 9
Cataract (Eye disorders) | 8 | 4 | 6
Nasopharyngitis (Infections and infestations) | 7 | 6 | 5
Intraocular pressure increased (Investigations) | 3 | 7 | 10

LIMITATIONS AND CAVEATS:
Study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No